CLINICAL TRIAL: NCT03490279
Title: Symptomatic Uncomplicated Diverticular Disease: a lactofErriN piLot studY
Brief Title: Lactoferrin for the Treatment of Symptomatic Uncomplicated Diverticular Disease
Acronym: SUDDENLY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Antonio Di Sabatino, Full Professor of Internal Medicine, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SUDDENLY17
Record Dates: First submitted 2018-03-30; First posted 2018-04-06 (Actual); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Diverticular Disease; Symptomatic Uncomplicated Diverticular Disease
MeSH Terms: conditions — Diverticular Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (Experimental): Lactoferrin CRX 100 mg, capsule formulation, 2 tablets taken together once daily, on an empty stomach (before breakfast)
  Interventions: Dietary Supplement: Lactoferrin CRX
- B (Placebo Comparator): Placebo 100 mg, capsule formulation, 2 tablets taken together once daily, on an empty stomach (before breakfast)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Lactoferrin CRX — Patients will be asked to take lactoferrin CRX as already mentioned (blindly).
  Arms: A
Other: Placebo — Patients will be asked to take placebo as already mentioned (blindly).
  Arms: B

SUMMARY:
Diverticular disease is a chronic pathology, characterized by recurrent abdominal symptoms and a high social impact, with a high prevalence in developed countries, especially among the elderly. Diverticula are thought to develop from age-related degeneration of the mucosal wall and segmental increases in colon pressure resulting in bulging at points of weakness, typically at the insertion of the vasa recta. Classification of diverticular disease is largely based on symptoms: it begins with the development of diverticulosis, to asymptomatic disease, to symptomatic uncomplicated diverticular disease (SUDD) and finally to complicated disease when patients develop abscesses, phlegmon, bleeding, fistula and sepsis. Approximately the 20% of the patients with diverticular disease has symptoms, such as abdominal pain, fever and altered bowel movement and, in the last decades, a significant increase of the incidence of complications related to the disease has been recorded, in particular of intestinal perforation.

Lactoferrin (Lf) is a glycoprotein present in several secretory liquids - i.e. milk, saliva and tears - with antimicrobial properties that it exert to seizing iron, thus preventing the use by the pathogens, or altering their plasma membrane through its highly cationic charge.

The investigators hypothesize that the antimicrobial and immunoregulatory characteristics of the Lf can be used to maintain an adequate homeostasis of the intestinal mucosa in patients with SUDD resulting in an improvement of both symptoms and quality of life.

DETAILED DESCRIPTION:
The investigators will verify whether a 4-week treatment with lactoferrin CRX is able to reduce SUDD-related symptoms, thus improving patient's quality of life. Symptoms will be assessed with the questionnaire by Tursi et al.

ELIGIBILITY:
Inclusion Criteria:

To be included in the trial the patient must:

* Have given written informed consent to participate
* Age ≥18 and <65 years
* Diagnosis of SUDD deﬁned as the presence of symptoms (mainly abdominal pain, but also constipation, diarrhoea and bloating) in patients with a previous diagnosis of diverticular disease at colonoscopy or imaging in the absence of any current complication (stenoses, abscesses, ﬁstulas)
* Women of childbearing potential are required to have a negative pregnancy test at the Baseline Visit (V1) and to use adequate contraception for the duration of the trial and for 14 days after the completion of the trial/last treatment. This includes:

  * Intrauterine Device
  * Hormonal based contraception (pill, contraceptive injection or implant etc)
  * Barrier contraception (condom and occlusive cap e.g. diaphragm or cervical cap with spermicide)
  * True abstinence (where this is in accordance with the patients preferred and usual lifestyle)
* Men are required to use adequate contraception for the entire duration of the trial and for 14 days after the completion of the trial/last treatment. This includes:

  * Barrier contraception (condom and spermicide) even if female partner(s) are using another method of contraception or are already pregnant (also to protect male partners from exposure to the trial product)
  * True abstinence (where this is in accordance with the patients preferred and usual lifestyle)

Exclusion Criteria:

The presence of any of the following will preclude patient inclusion:

* Patients diagnosed with irritable bowel syndrome, bacterial and/or parasitic intestinal diseases, inflammatory bowel disease
* Female patients who are pregnant or breastfeeding
* Use of the following medications:

  1. Use of oral or rectal 5-aminosalicylic (5-ASA) 7 days prior to enrollment
  2. Use of antibiotics for diverticular disease within the 7 days prior to enrollment
  3. Use of probiotics within the 7 days prior to enrollment
* Known history of drug or alcohol abuse within the last 3 years prior to enrollment
* Any unstable or uncontrolled cardiovascular, pulmonary, hepatic, renal, gastrointestinal, genitourinary, hematological, coagulation, immunological, endocrine/metabolic, or other medical disorder that, in the opinion of the investigator, would confound the study results or compromise patient safety
* Any surgical procedure requiring general anesthesia within 30 days prior to enrollment or is planning to undergo major surgery during the study period
* Active participation in other interventional or drug research in the study period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-05-02 (Estimated); Study Completion 2019-11-02 (Estimated)

PRIMARY OUTCOMES:
Abdominal symptoms reduction | 4 weeks
  The primary outcome measure is the percentage of patients with a reduction of at least the 50% of the symptoms according to the Tursi questionnaire.

SECONDARY OUTCOMES:
Symptom-free remission | 4 week
  The percentage of patients that will achieve symptom-free remission after a 4-week course of lactoferrin CRX vs placebo, according to the Tursi questionnaire.
36-item short form survey (SF-36) | 4 weeks
  Evaluation of the quality of life after a 4-week course of lactoferrin CRX vs placebo, according to the 36-item short form survey (SF-36)
Fecal microbiota | 4 weeks
  Evaluation of fecal microbiota after a 4-week course of lactoferrin CRX vs placebo

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, Pavia, Italy

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD), anonymized and aggregated, that underlie results in a publication.
Supporting Information: SAP, CSR
Time Frame: Only on future articles that will be published.